CLINICAL TRIAL: NCT03506763
Title: Effect of Pre-medication in Pain Measures on Office Hysteroscopy - Randomized Clinical Trial
Brief Title: Effect of Pre-medication in Pain Measures on Office Hysteroscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 65409017.0.0000.5327
Record Dates: First submitted 2018-04-13; First posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Pain
Keywords: office hysteroscopy, pain measure
MeSH Terms: conditions — Pain | interventions — Diclofenac; Tablets

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider, Investigator
Masking Description: RCT, blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo Oral + Placebo Oral (Placebo Comparator): Placebo Oral + Placebo Oral
  Interventions: Drug: Placebo Oral + Placebo Oral
- Diclofenac oral + Placebo Oral (Active Comparator): Diclofenac oral + Placebo Oral
  Interventions: Drug: Diclofenac oral + Placebo Oral
- Diclofenac oral + scopolamina oral (Active Comparator): Diclofenac oral + scopolamina oral
  Interventions: Drug: Diclofenac oral + scopolamina oral

INTERVENTIONS:
Drug: Placebo Oral + Placebo Oral — Placebo Oral + Placebo Oral
  Other Names: Placebo
  Arms: Placebo Oral + Placebo Oral
Drug: Diclofenac oral + Placebo Oral — Diclofenac oral + Placebo Oral
  Other Names: Diclofenac 50 mg oral tablet
  Arms: Diclofenac oral + Placebo Oral
Drug: Diclofenac oral + scopolamina oral — Diclofenac oral + scopolamina oral
  Other Names: Diclofenac 50 mg oral tablet, scopolamin 10 mg oral tablet
  Arms: Diclofenac oral + scopolamina oral

SUMMARY:
Will be perform a RCT to compare pain measure on office hysteroscopy after pre-medication with oral analgesic. Patients will be alocate to oral sodic diclofenac, scopolamin or placebo. We will compare visual analog score of pain after the procedure.

Patients: patients with indication of office hysteroscopy to evaluate uterine intracavitary abnormality.

Interventions Group 1 (control) The patients will receive about 2 h prior to the procedure 2 placebo tablets.

Group 2 (diclofenac + scopolamine) The patients will receive about 2 h prior to the procedure 1 tablet of diclofenac sodium 50 mg and 1 tablet of scopolamine 2 mg.

Group 3 (diclofenac only). Patients will receive approximately 2 h prior to the procedure 1 tablet of diclofenac sodium 50 mg and 1 tablet of placebo.

DETAILED DESCRIPTION:
Pain during and 30 minutes after a hysteroscopy will be measured through the visual analog pain scale of 10 centimeters, considering 0 (no pain) and 10 (unbearable pain or the greatest pain ever experienced). Acceptance of the procedure and assessed through the Likert 5-point scale: 1) totally disagree; 2) disagree; 3) I do not agree or disagree; 4) I agree and 5) I totally agree.There will also be a need for analgesia after the procedure, the time spent in the observation room and the onset of vagal symptoms such as dizziness, malaise, nausea, vomiting or syncope

ELIGIBILITY:
Inclusion Criteria:

1. indication of intrauterine evaluation
2. Abnormal uterine bleeding
3. post-menopause uterine bleeding
4. infertility
5. recurrent miscarriage

Exclusion Criteria:

1. stenosis of the external cervical orifice,
2. pelvic inflammatory disease,
3. suspected gestation or pregnancy,
4. active bleeding at the time of examination
5. contraindication to the use of the study medication, diclofenac sodium and scopolamine,

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain measure | until 1 hour after exam
  Pain Visual analogue score

SECONDARY OUTCOMES:
Likert scale | until 1 hour after exam
  Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Joao Sabino, MD, Principal Investigator — HCPA- Professor
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided